CLINICAL TRIAL: NCT04609553
Title: Addressing Disparities in Language and Social-emotional Skill Acquisition Through Literacy Promotion in Primary Care: Literacy Promotion for Latinos Study
Brief Title: Literacy Promotion for Latinos Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Manuel E. Jimenez, MD, MS, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro2019002784; 1R01HD099125-01A1 (NIH)
Record Dates: First submitted 2020-10-21; First posted 2020-10-30 (Actual); Results first posted 2025-11-25 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Language Development; Behavior, Child; Parenting; Literacy
Keywords: literacy promotion, early childhood, Latino, primary care
MeSH Terms: conditions — Child Behavior; Literacy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care including ROR (Active Comparator): Literacy promotion is a pediatric standard of care. Participants in this group will receive usual care that includes ROR, a primary care literacy promotion intervention.
  Interventions: Behavioral: Usual care including ROR
- ROR plus text messages (Experimental): In addition to ROR, participants will receive three text messages per week, plus one interactive follow-up message per month, for the study period with scheduled breaks.
  Interventions: Behavioral: Usual care including ROR; Behavioral: Text messages
- ROR plus text messages plus connection to community resources (Experimental): In addition to ROR and text messages, participants will be referred to a county-based single point of entry system for referrals to community resources. This system simplifies access to poverty-reducing resources by creating a centralized access point, maintaining an updated data base of resources with existing capacity to support families, and providing case management.
  Interventions: Behavioral: Usual care including ROR; Behavioral: Text messages; Behavioral: Connection to community resources

INTERVENTIONS:
Behavioral: Usual care including ROR — Usual care which includes ROR.
Behavioral: Text messages — 3 text messages per week and one interactive text per month.
  Arms: ROR plus text messages; ROR plus text messages plus connection to community resources
Behavioral: Connection to community resources — Referral to a non-profit that connects families with community resources and provides families with case management.
  Arms: ROR plus text messages plus connection to community resources

SUMMARY:
This study tests the extent to which tailored outreach text messages that provide a cue to action and an intervention that enhances access to poverty-reducing resources, in combination with standard primary care literacy promotion, can improve child language and social- emotional skill acquisition among low-income Latino children.

DETAILED DESCRIPTION:
The investigators propose a 3 arm randomized clinical trial to test strategies designed to enhance literacy promotion for low-income Latino families. The investigators will recruit 630 parent-child dyads from community health centers that serve low-income, Latino families. Parents will be randomly assigned to one of 3 arms (1) Reach Out and Read (ROR) an evidence-based literacy promotion intervention that is widely disseminated in primary care; (2) ROR plus tailored outreach text messages; (3) ROR plus tailored outreach text messages and enhanced access to poverty-reducing resources using a widely disseminated model that simplifies access and provides care coordination. In Aim 1, the investigators will test their hypotheses that (1) children in the ROR plus text message arm will have higher scores on validated assessments of language and social-emotional development compared to standard ROR alone and (2) children who receive both text messages and enhanced access to poverty-reducing resources will have higher scores compared to the other two arms. In Aim 2, the investigators will examine mechanisms that underlie the effects of the interventions. In Aim 3, the investigators will use mixed methods to conduct a process evaluation to understand how the interventions are implemented, identify barriers, facilitators, and modifications, and explore parents' experiences with the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregiver of a child age 6 months to 12 months
* Identifies as Latino/a/x
* Primary language English or Spanish
* Cell phone ownership
* Age 18 years or older
* Willing to receive text messages
* Willing to accept being placed into one of three study groups

Exclusion Criteria:

* Children with multiple congenital anomalies or genetic disorders and previously identified developmental delays
* Individuals unable to provide informed consent
* Intent to discontinue care at current pediatric clinic / recruitment site
* Discontinued care at one of the three pediatric clinics / recruitment sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 662 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2024-12-28 (Actual); Study Completion 2024-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel E Jimenez, MD, MS, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified quantitative data and associated documentation may be made available to users conducting non-profit research under a written data-sharing agreement.
Supporting Information: Study Protocol
Time Frame: Data will become available after the study is completed and primary study findings are published in peer-reviewed journals.
Access Criteria: Researchers from accredited institutions may request access to the data for non-profit research. Permission and access will be granted on an ad hoc basis. Only deidentified data will be made available.

REFERENCES:
- [Derived] Zanzoul S, Strickland PO, Mendelsohn AL, Malke K, Bator A, Hemler J, Jimenez ME. Stress and Infant Media Exposure During COVID-19: A Study Among Latino Families. J Dev Behav Pediatr. 2024 Jan 1;45(1):e14-e20. doi: 10.1097/DBP.0000000000001231. Epub 2023 Dec 21. PMID 38127845

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from three health centers in central New Jersey between November 2020 and June 2023.
Pre-assignment Details: 1,129 potential participants were assessed for eligibility, and of these, 467 were excluded, and 662 met inclusion criteria and were consented. Of these 662 participants, 630 were randomized. Of the other 32 who were not randomized, 17 declined to participate and 15 lost contact.
Groups:
- Usual care including ROR: Literacy promotion is a pediatric standard of care. Participants in this group received usual care that includes ROR, a primary care literacy promotion intervention.
  Usual care including ROR: Usual care which includes ROR.
- ROR plus text messages: In addition to ROR, participants received three text messages per week, plus one interactive follow-up message per month, for the study period with scheduled breaks.
  Usual care including ROR: Usual care which includes ROR.
  Text messages: 3 text messages per week and one interactive text per month.
- ROR plus text messages plus connection to community resources: In addition to ROR and text messages, participants were referred to a county-based single point of entry system for referrals to community resources. This system simplifies access to poverty-reducing resources by creating a centralized access point, maintaining an updated data base of resources with existing capacity to support families, and providing case management.
  Usual care including ROR: Usual care which includes ROR.
  Text messages: 3 text messages per week and one interactive text per month.
  Connection to community resources: Referral to a non-profit that connects families with community resources and provides families with case management.
Period: Overall Study
Arm/Group | Usual care including ROR | ROR plus text messages | ROR plus text messages plus connection to community resources
Started | 209 (This number reflects the number of caregiver/child dyads in arm 1 who began the study. Thus, there were 209 unique caregivers and 209 unique children in arm 1 who started the study.) | 210 (This number reflects the number of caregiver/child dyads in arm 2 who began the study. Thus, there were 210 unique caregivers and 210 unique children in arm 2 who started the study.) | 211 (This number reflects the number of caregiver/child dyads in arm 3 who began the study. Thus, there were 211 unique caregivers and 211 unique children in arm 3 who started the study.)
9-month follow up | 168 (This number reflects the number of caregiver/child dyads in arm 1 who completed the 9-month follow-up. Thus, there were 168 unique caregivers and 168 unique children in arm 1 who participated in the 9-month follow-up.) | 173 (This number reflects the number of caregiver/child dyads in arm 2 who completed the 9-month follow-up. Thus, there were 173 unique caregivers and 173 unique children in arm 2 who participated in the 9-month follow-up.) | 178 (This number reflects the number of caregiver/child dyads in arm 3 who completed the 9-month follow-up. Thus, there were 178 unique caregivers and 178 unique children in arm 3 who participated in the 9-month follow-up.)
Completed | 170 (This number reflects the number of caregiver/child dyads in arm 1 who completed the study. Thus, there were 170 unique caregivers and 170 unique children in arm 1 who completed the study.) | 169 (This number reflects the number of caregiver/child dyads in arm 2 who completed the study. Thus, there were 169 unique caregivers and 169 unique children in arm 2 who completed the study.) | 178 (This number reflects the number of caregiver/child dyads in arm 3 who completed the study. Thus, there were 178 unique caregivers and 178 unique children in arm 3 who completed the study.)
Not Completed | 39 | 41 | 33
Not completed — Lost to Follow-up | 27 | 31 | 24
Not completed — Discontinued | 12 | 10 | 9

BASELINE CHARACTERISTICS:
Population: The overall number of baseline participants represents the number of caregiver/child dyads in each arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care Including ROR | ROR Plus Text Messages | ROR Plus Text Messages Plus Connection to Community Resources | Total
Number analyzed (Participants) | 209 | 210 | 211 | 630
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of the caregiver in the caregiver/child dyad.
  years | 30.4 (6.4) | 31.5 (6.7) | 30.7 (5.9) | 31.0 (6.3)
Age, Continuous [Mean (Standard Deviation); unit: months] — Age of the child in the caregiver/child dyad.
  months | 7.8 (1.4) | 8.0 (1.5) | 8.1 (1.5) | 8.0 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex of the caregiver in the caregiver/child dyad.
  Participants
    Female | 205 | 207 | 204 | 616
    Male | 4 | 3 | 7 | 14
Sex: Female, Male [Count of Participants; unit: Participants] — Sex of the child in the caregiver/child dyad.
  Participants
    Female | 92 | 110 | 117 | 319
    Male | 117 | 100 | 94 | 311
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — All participants self-identified as Latino/a/x as this was part of the inclusion criteria.
  Participants
    Hispanic or Latino | 209 | 210 | 211 | 630
    Not Hispanic or Latino | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Caregiver's Self-reported Rating of Ability to Speak English [Count of Participants; unit: Participants]
  Speaks Very Well | 25 | 25 | 27 | 77
  Speaks Well | 29 | 51 | 29 | 109
  Speaks Not Well | 78 | 71 | 81 | 230
  Speaks Not at All | 76 | 62 | 74 | 212
  Missing | 1 | 1 | 0 | 2
Caregiver's Highest Level of Education [Count of Participants; unit: Participants]
  < High School | 35 | 33 | 36 | 104
  Some High School | 40 | 29 | 41 | 110
  High School Graduate | 80 | 95 | 75 | 250
  Some College | 26 | 26 | 25 | 77
  ≥ College graduate | 28 | 26 | 34 | 88
  Missing | 0 | 1 | 0 | 1
Caregiver Health Literacy Score [Mean (Standard Deviation); unit: units on a scale] — Health literacy score was assessed using the Short Assessment of Health Literacy (SAHL), and was administered in English or Spanish, based on the participant's language preference. The SAHL has 18 questions, with each question including (1) correctly reading a health-related word aloud, and (2) hearing 2 additional words, and choosing the one most closely related to the original health-related word.
  Total possible scores range from 0-18, with scores 14 and below indicating low health literacy.
  units on a scale | 15.7 (2.7) | 15.4 (2.8) | 15.9 (1.8) | 15.7 (2.5)
Child Social-Emotional Skills [Mean (Standard Deviation); unit: T-score] — Child's social-emotional skills were assessed with the Devereux Early Childhood Assessment for Infants and Toddlers (DECA-I/T), which has 2 caregiver-report forms: an infant form (1-18 months) that includes Attachment/Relationships and Initiative subscales, and a toddler form (18-36 months) that includes Attachment/Relationships, Initiative, and Self-Regulation subscales. Scores are standardized on a T-distribution (M=50; SD=10). The Total Protective Factors score is calculated by adding subscale T-scores. T-scores of 60+ indicate an area strength, and T-scores of 40- indicate an area need.
  T-score | 95.7 (18.3) | 93.8 (17.8) | 94.5 (18.3) | 94.7 (18.2)
Reading Activities [Mean (Standard Deviation); unit: units on a scale] — Reading activities were assessed with the STIMQ2 reading scale, a parent-report measure. Subscales include Quantity, Diversity, and Quality. Total possible scores range from 0 to 19, with higher scores equating to higher quantity, diversity, and quality of shared reading.
  units on a scale | 4.5 (3.9) | 4.0 (3.9) | 4.2 (3.9) | 4.2 (3.9)
Community Resource Participation [Mean (Standard Deviation); unit: units on a scale] — Community resource participation was measures via the Survey of Income and Program Participation (SIPP), a self-reported measure of participation in different types of community resources (e.g., food/nutrition support, income support, childcare assistance, etc.). Possible scores range from 0 to 17, with higher scores indicating more involvement in community resources.
  units on a scale | 2.6 (1.2) | 2.5 (1.2) | 2.7 (1.2) | 2.6 (1.2)
Caregiver-Clinician Relationship [Mean (Standard Deviation); unit: units on a scale] — Caregiver-clinician relationship was assessed with the Modified Physician-Parent Communication Survey, Interest subscale. The interest subscale includes 6 items scored from 1 to 8. Item scores are then averaged. Total possible scores range from 1-8, with higher scores indicating stronger relationships.
  units on a scale | 5.8 (1.9) | 5.7 (1.9) | 5.5 (2.1) | 5.7 (1.9)
Economic Stress [Mean (Standard Deviation); unit: units on a scale] — Economic stress was assessed using the Local Inventory of Needs and Knowledge (LINK). Questions are answered on a 5-point Likert scale of "strongly disagree" (0) to "strongly agree" (4). Possible scores range from 0 to 16 with higher scores indicating greater needs and economic stress.
  units on a scale | 2.6 (1.1) | 2.7 (2.0) | 2.7 (1.1) | 2.7 (1.1)
Parent Stress [Mean (Standard Deviation); unit: units on a scale] — Caregiver stress was measured via the Parental Stress Scale (PSS), an 18-item scale. For each item, parents rate how much they agree or disagree using a 5-point Likert scale ranging from "strongly disagree" (1) to "strongly agree" (5). Total possible scores range from 18 to 90 with higher scores indicating more parental stress.
  units on a scale | 34.4 (7.9) | 35.1 (7.8) | 34.8 (7.5) | 34.8 (7.7)
Child Media Use [Mean (Standard Deviation); unit: units on a scale] — Child media use was measured using the Modified ScreenQ-I/T 2.0 (Infant/Toddler) version. There are 15 items, with total possible scores ranging from 0 to 26. Higher scores indicate more child media use.
  units on a scale | 4.9 (3.2) | 4.7 (2.7) | 4.6 (2.9) | 4.7 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Child Language Skills
Description: Expressive One-Word Picture Vocabulary Test - Fourth Edition (EOWPVT-4) Spanish-Bilingual - Assesses expressive language skills in English and Spanish. This multiple-choice format test consists of 190 items presented in developmental sequence; age-related starting points and cut-off points ensure that only a subset of items is administered. Raw scores are converted into standard scores (M=100, SD=15). Higher scores denote stronger language skills, with possible standard scores ranging between 55 and 145.
Time Frame: 18-month follow-up
Population: Participants include those who had baseline data and completed the EOWPVT at the 18-month follow-up. The EOWPVT was only administered at the 18-month follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual care including ROR | ROR plus text messages | ROR plus text messages plus connection to community resources
Number analyzed (Participants) | 168 | 163 | 173
score on a scale | 2.1 (4.2) | 2.3 (4.2) | 2.6 (4.4)
Statistical Analysis 1: Comparison: Usual care including ROR vs ROR plus text messages; A total of 630 parent-infant dyads (210 per arm) were needed to achieve 80% power to detect a 0.3 standard deviation (SD) difference assuming approximately 20% attrition. The null hypothesis was that there would be no differences between Arm 1 and Arm 2; Test type: Superiority; p = 0.64, ANOVA — p-value is adjusted using the minP approach for potentially highly correlated outcomes. Then, p < 0.05 was used as an a priori threshold for statistical significance; We followed the intent to treat principle, with participants included based on their group assignment. Because of the multiple, potentially highly correlated primary outcomes, we used the step-down minP method (a re-sampling approach), to assess the effects of treatment across primary outcomes and timepoints within domain (total=3 outcomes within the language development). Right skewed variables with minimum values of zero were log-transformed after adding one. minP-adjusted p-values were calculated with ANOVA models comparing outcomes adjusted for correlations due to repeated-measure effects for both active treatments versus control. Specifically, no adjustments were made for child expressive language since it was only measured at 18 months
Statistical Analysis 2: Comparison: Usual care including ROR vs ROR plus text messages plus connection to community resources; A total of 630 parent-infant dyads (210 per arm) were needed to achieve 80% power to detect a 0.3 standard deviation (SD) difference assuming approximately 20% attrition. The null hypothesis was that there would be no differences between Arm 1 and Arm 3; Test type: Superiority; p = 0.46, ANOVA — [p-value comment as in outcome 1, analysis 1]; [other analysis details as in outcome 1, analysis 1]

2. Primary Outcome: Child Communicative Skills
Description: Caregiver report of non-verbal communication and early expressive language assessed using the MacArthur Bates Communicative Development Inventories. The Words & Gestures short form is an 89-word vocabulary checklist with separate columns for comprehension and production for children 8-18 months. The Words & Sentences versions contain a 100-word productive vocabulary checklist and a question about combining words for children 16-30 months. Scores are summed and higher scores denote stronger skills.
Time Frame: 9-month follow-up, 18-month follow-up
Population: Analyses for the 9-month and 18-month follow-up visits include participants who had baseline data and completed the MacArthur Bates Communicative Development Inventories at the 9-month and/or 18-month follow-up visit(s), respectively. Participants who did not participate in the 9-month follow-up were still welcome to participate in the 18-month follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual care including ROR | ROR plus text messages | ROR plus text messages plus connection to community resources
Number analyzed (Participants) | 194 | 193 | 201
score on a scale
  9-month follow-up: number analyzed (Participants) | 168 | 173 | 178
  9-month follow-up | 12.5 (13.7) | 13.5 (14.4) | 15.7 (20.9)
  18-month follow-up: number analyzed (Participants) | 170 | 169 | 178
  18-month follow-up | 44.5 (32.2) | 50.4 (30.8) | 46.6 (32.1)
Statistical Analysis 1: Comparison: Usual care including ROR vs ROR plus text messages; Analysis for 9-month follow-up. A total of 630 parent-infant dyads (210 per arm) were needed to achieve 80% power to detect a 0.3 standard deviation (SD) difference assuming approximately 20% attrition. The null hypothesis was that there would be no differences between Arm 1 and Arm 2; Test type: Superiority; p = 0.84, ANOVA — [p-value comment as in outcome 1, analysis 1]; We followed the intent to treat principle, with participants included based on their group assignment. Because of the multiple, potentially highly correlated primary outcomes, we used the step-down minP method (a re-sampling approach), to assess the effects of treatment across primary outcomes and timepoints within domain (total=3 outcomes within the language development). Right skewed variables with minimum values of zero were log-transformed after adding one. minP-adjusted p-values were calculated with ANOVA models comparing outcomes adjusted for correlations due to repeated-measure effects for both active treatments versus control. The adjusted value for child communicative development was the value of the outcome minus the best linear unbiased predictor (BLUP) estimated from a mixed linear model with random individual-specific intercepts and treatment fixed effects
Statistical Analysis 2: Comparison: Usual care including ROR vs ROR plus text messages plus connection to community resources; Analysis for 9-month follow-up. A total of 630 parent-infant dyads (210 per arm) were needed to achieve 80% power to detect a 0.3 standard deviation (SD) difference assuming approximately 20% attrition. The null hypothesis was that there would be no differences between Arm 1 and Arm 3; Test type: Superiority; p = 0.82, ANOVA — [p-value comment as in outcome 1, analysis 1]; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Usual care including ROR vs ROR plus text messages; Analysis for 18-month follow-up. A total of 630 parent-infant dyads (210 per arm) were needed to achieve 80% power to detect a 0.3 standard deviation (SD) difference assuming approximately 20% attrition. The null hypothesis was that there would be no differences between Arm 1 and Arm 2; Test type: Superiority; p = 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Usual care including ROR vs ROR plus text messages plus connection to community resources; Analysis for 18-month follow-up. A total of 630 parent-infant dyads (210 per arm) were needed to achieve 80% power to detect a 0.3 standard deviation (SD) difference assuming approximately 20% attrition. The null hypothesis was that there would be no differences between Arm 1 and Arm 3; Test type: Superiority; p = 0.16, ANOVA — [p-value comment as in outcome 1, analysis 1]; [other analysis details as in outcome 2, analysis 1]

3. Primary Outcome: Child Social-emotional Skills
Description: Child's social-emotional skills were assessed with the Devereux Early Childhood Assessment for Infants and Toddlers (DECA-I/T), which has 2 caregiver-report forms: an infant form (1-18 months) that includes Attachment/Relationships and Initiative subscales, and a toddler form (18-36 months) that includes Attachment/Relationships, Initiative, and Self-Regulation subscales. Scores are standardized on a T-distribution (M=50; SD=10). The Total Protective Factors score is calculated by adding subscale T-scores. T-scores of 60+ indicate an area strength, and T-scores of 40- indicate an area need.
Time Frame: Baseline, 9-month follow-up, 18-month follow-up
Population: Analyses for the 9-month and 18-month follow-up visits include participants who had baseline data and completed the DECA at the 9-month and/or 18-month follow-up visit(s), respectively. Participants who did not participate in the 9-month follow-up were still welcome to participate in the 18-month follow-up.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Usual care including ROR | ROR plus text messages | ROR plus text messages plus connection to community resources
Number analyzed (Participants) | 207 | 208 | 209
T-score
  Baseline | 95.7 (18.3) | 93.8 (17.8) | 94.5 (18.3)
  9-month follow-up: number analyzed (Participants) | 168 | 171 | 176
  9-month follow-up | 88.4 (17.2) | 87.9 (19.2) | 91.4 (18.9)
  18-month follow-up: number analyzed (Participants) | 170 | 166 | 177
  18-month follow-up | 133.5 (26.5) | 138.4 (28.4) | 140.6 (24.6)
Statistical Analysis 1: Comparison: Usual care including ROR vs ROR plus text messages; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.93, ANOVA — [p-value comment as in outcome 1, analysis 1]; We followed the intent to treat principle, with participants included based on their group assignment. Because of the multiple correlated timepoints within the social emotional domain, we used the step-down minP method (a re-sampling approach), to assess the effects of treatment (total=2 outcomes within the social emotional). minP-adjusted p-values were calculated with ANOVA models comparing outcomes adjusted for baseline- and correlations due to repeated-measure effects for both active treatments versus control. The adjusted value for social emotional development was the value of the outcome minus the effect of baseline and the best linear unbiased predictor (BLUP) estimated from a mixed linear model with random individual-specific intercepts and both treatment and baseline fixed effects
Statistical Analysis 2: Comparison: Usual care including ROR vs ROR plus text messages plus connection to community resources; Analysis for 9-month follow-up, A total of 630 parent-infant dyads (210 per arm) were needed to achieve 80% power to detect a 0.3 standard deviation (SD) difference assuming approximately 20% attrition. The null hypothesis was that there would be no differences between Arm 1 and Arm 3; Test type: Superiority; p = 0.04, ANOVA — [p-value comment as in outcome 1, analysis 1]; [other analysis details as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Usual care including ROR vs ROR plus text messages; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.08, ANOVA — [p-value comment as in outcome 1, analysis 1]; [other analysis details as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Usual care including ROR vs ROR plus text messages plus connection to community resources; [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p = 0.03, ANOVA — [p-value comment as in outcome 1, analysis 1]; [other analysis details as in outcome 3, analysis 1]

4. Primary Outcome: Caregiver Cognitive Stimulation
Description: The StimQ2 is a caregiver-reported measure of cognitive stimulation for children that includes domains on the home literacy environment (Reading scale) and responsiveness (Parental Verbal Responsiveness scale). The Reading scale includes 3 subdimensions (Book Reading Quantity, Diversity of Content, Book Reading Quality). Scores on the Reading scale range from 0 to 19. The Parental Verbal Responsiveness scale is composed of two subdimensions (Everyday Routines and Play and Pretend). Scores range from 0 to 15. Higher scores indicate more cognitive stimulation. The Reading scale was completed at baseline, the 9-month follow-up, and the 18-month follow-up. The Parent Verbal Responsiveness scale was completed at the 9-month follow-up and the18-month follow-up.
Time Frame: Baseline, 9-month follow-up, 18-month follow-up
Population: Analyses for the 9-month and 18-month follow-up visits include participants who had baseline data and completed the StimQ2 at the 9-month and/or 18-month follow-up visit(s), respectively. Participants who did not participate in the 9-month follow-up were still welcome to participate in the 18-month follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual care including ROR | ROR plus text messages | ROR plus text messages plus connection to community resources
Number analyzed (Participants) | 209 | 210 | 211
score on a scale
  Baseline (Reading) | 4.5 (3.9) | 4.0 (3.9) | 4.2 (3.9)
  9-month follow-up (Reading): number analyzed (Participants) | 168 | 173 | 178
  9-month follow-up (Reading) | 6.0 (3.8) | 6.7 (3.5) | 6.1 (3.8)
  18-month follow-up (Reading): number analyzed (Participants) | 170 | 168 | 178
  18-month follow-up (Reading) | 6.6 (4.2) | 6.8 (4.0) | 6.7 (4.1)
  9-month follow-up (Parent Verbal Responsiveness): number analyzed (Participants) | 168 | 172 | 178
  9-month follow-up (Parent Verbal Responsiveness) | 5.5 (2.3) | 5.8 (2.1) | 6.1 (2.0)
  18-month follow-up (Parent Verbal Responsiveness): number analyzed (Participants) | 169 | 168 | 178
  18-month follow-up (Parent Verbal Responsiveness) | 6.5 (1.9) | 6.4 (2.1) | 6.8 (1.9)
Statistical Analysis 1: Comparison: Usual care including ROR vs ROR plus text messages; Analysis for the Reading Scale at the 9-month follow-up. A total of 630 parent-infant dyads (210 per arm) were needed to achieve 80% power to detect a 0.3 standard deviation (SD) difference assuming approximately 20% attrition. The null hypothesis was that there would be no differences between Arm 1 and Arm 2; Test type: Superiority; p = 0.002, ANOVA — [p-value comment as in outcome 1, analysis 1]; We followed the intent to treat principle, with participants included based on their group assignment. Because of the multiple correlated timepoints within the parental behavior domain, we used the step-down minP method (a re-sampling approach), to assess the effects of treatment (total=6 outcomes within the parental behavior). minP-adjusted p-values were calculated with ANOVA models comparing outcomes adjusted for baseline- and correlations due to repeated-measure effects (as appropriate) for both active treatments versus control. The adjusted value for reading activities was the value of the outcome minus the effect of baseline and the best linear unbiased predictor (BLUP) estimated from a mixed linear model with random individual-specific intercepts and both treatment and baseline fixed effects
Statistical Analysis 2: Comparison: Usual care including ROR vs ROR plus text messages plus connection to community resources; Analysis for the Reading Scale at the 9-month follow-up. A total of 630 parent-infant dyads (210 per arm) were needed to achieve 80% power to detect a 0.3 standard deviation (SD) difference assuming approximately 20% attrition. The null hypothesis was that there would be no differences between Arm 1 and Arm 3; Test type: Superiority; p = 0.80, ANOVA — [p-value comment as in outcome 1, analysis 1]; [other analysis details as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Usual care including ROR vs ROR plus text messages; Analysis for the Reading Scale at the18-month follow-up. A total of 630 parent-infant dyads (210 per arm) were needed to achieve 80% power to detect a 0.3 standard deviation (SD) difference assuming approximately 20% attrition. The null hypothesis was that there would be no differences between Arm 1 and Arm 2; Test type: Superiority; p = 0.79, ANOVA — [p-value comment as in outcome 1, analysis 1]; [other analysis details as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Usual care including ROR vs ROR plus text messages plus connection to community resources; Analysis for the Reading Scale at the 18-month follow-up. A total of 630 parent-infant dyads (210 per arm) were needed to achieve 80% power to detect a 0.3 standard deviation (SD) difference assuming approximately 20% attrition. The null hypothesis was that there would be no differences between Arm 1 and Arm 3; Test type: Superiority; p = 0.96, ANOVA — [p-value comment as in outcome 1, analysis 1]; [other analysis details as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Usual care including ROR vs ROR plus text messages; Analysis for the Parent Verbal Responsiveness Scale at the 9-month follow-up. A total of 630 parent-infant dyads (210 per arm) were needed to achieve 80% power to detect a 0.3 standard deviation (SD) difference assuming approximately 20% attrition. The null hypothesis was that there would be no differences between Arm 1 and Arm 2; Test type: Superiority; p = 0.22, ANOVA — [p-value comment as in outcome 1, analysis 1]; We followed the intent to treat principle, with participants included based on their group assignment. Because of the multiple correlated timepoints within the parental behavior domain, we used the step-down minP method (a re-sampling approach), to assess the effects of treatment (total=6 outcomes within the parental behavior). minP-adjusted p-values were calculated with ANOVA models comparing outcomes adjusted for baseline- and correlations due to repeated-measure effects (as appropriate) for both active treatments versus control. The adjusted value for verbal responsiveness was the value of the outcome minus the best linear unbiased predictor (BLUP) estimated from a mixed linear model with random individual-specific intercepts and treatment fixed effects
Statistical Analysis 6: Comparison: Usual care including ROR vs ROR plus text messages plus connection to community resources; Analysis for the Parent Verbal Responsiveness Scale at the 9-month follow-up. A total of 630 parent-infant dyads (210 per arm) were needed to achieve 80% power to detect a 0.3 standard deviation (SD) difference assuming approximately 20% attrition. The null hypothesis was that there would be no differences between Arm 1 and Arm 3; Test type: Superiority; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; [other analysis details as in outcome 4, analysis 5]
Statistical Analysis 7: Comparison: Usual care including ROR vs ROR plus text messages; Analysis for the Parent Verbal Responsiveness Scale at the 18-month follow-up. A total of 630 parent-infant dyads (210 per arm) were needed to achieve 80% power to detect a 0.3 standard deviation (SD) difference assuming approximately 20% attrition. The null hypothesis was that there would be no differences between Arm 1 and Arm 2; Test type: Superiority; p = 0.96, ANOVA — [p-value comment as in outcome 1, analysis 1]; [other analysis details as in outcome 4, analysis 5]
Statistical Analysis 8: Comparison: Usual care including ROR vs ROR plus text messages plus connection to community resources; Analysis for the Parent Verbal Responsiveness Scale at the 18-month follow-up. A total of 630 parent-infant dyads (210 per arm) were needed to achieve 80% power to detect a 0.3 standard deviation (SD) difference assuming approximately 20% attrition. The null hypothesis was that there would be no differences between Arm 1 and Arm 3; Test type: Superiority; p = 0.12, ANOVA — [p-value comment as in outcome 1, analysis 1]; [other analysis details as in outcome 4, analysis 5]

5. Primary Outcome: Dialogic Reading Behavior
Description: The DialogPR is a caregiver report measure of shared reading quality. Score range from 0 to 30 with higher scores indicating more interactive reading.
Time Frame: 9-month follow-up
Population: Analyses for the 9-month visit include participants who had baseline data and completed the DialogPR at the 9-month visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual care including ROR | ROR plus text messages | ROR plus text messages plus connection to community resources
Number analyzed (Participants) | 168 | 171 | 178
score on a scale | 16.7 (10.0) | 18.1 (8.8) | 17.3 (10.1)
Statistical Analysis 1: Comparison: Usual care including ROR vs ROR plus text messages; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.78, ANOVA — [p-value comment as in outcome 1, analysis 1]; We followed the intent to treat principle, with participants included based on their group assignment. Because of the multiple correlated timepoints within the parental behavior domain, we used the step-down minP method (a re-sampling approach), to assess the effects of treatment (total=6 outcomes within the parental behavior). minP-adjusted p-values were calculated with ANOVA models comparing outcomes adjusted for baseline- and correlations due to repeated-measure effects (as appropriate) for both active treatments versus control. Dialogic reading behavior was measured at a single timepoint (9 months), so no adjustment was necessary
Statistical Analysis 2: Comparison: Usual care including ROR vs ROR plus text messages plus connection to community resources; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.96, ANOVA — [p-value comment as in outcome 1, analysis 1]; [other analysis details as in outcome 5, analysis 1]

6. Primary Outcome: Caregiver Discipline Strategies
Description: This questionnaire was modified from the National Survey of Early Childhood Health and asks two questions about verbal and physical discipline. Scores range from 0 to 6 and higher scores indicate harsher discipline strategies.
Time Frame: 18-month follow-up
Population: Analyses include participants who had baseline data and completed the caregiver discipline strategy measure at the 18-month follow-up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual care including ROR | ROR plus text messages | ROR plus text messages plus connection to community resources
Number analyzed (Participants) | 169 | 169 | 178
score on a scale | 1.9 (1.3) | 2.0 (1.4) | 2.1 (1.4)
Statistical Analysis 1: Comparison: Usual care including ROR vs ROR plus text messages; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.78, ANOVA — [p-value comment as in outcome 1, analysis 1]; We followed the intent to treat principle, with participants included based on their group assignment. Because of the multiple correlated timepoints within the parental behavior domain, we used the step-down minP method (a re-sampling approach), to assess the effects of treatment (total=6 outcomes within the parental behavior). minP-adjusted p-values were calculated with ANOVA models comparing outcomes adjusted for baseline- and correlations due to repeated-measure effects (as appropriate) for both active treatments versus control. Discipline strategies were measured at a single timepoint (18 months), so no adjustment was necessary
Statistical Analysis 2: Comparison: Usual care including ROR vs ROR plus text messages plus connection to community resources; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.96, ANOVA — [p-value comment as in outcome 1, analysis 1]; [other analysis details as in outcome 6, analysis 1]

7. Secondary Outcome: Caregiver Attitudes About Reading
Description: The Parent Reading Belief Inventory is a caregiver reported measure of attitudes about reading with children that included positive affect (scores range from 0 to 33). Higher scores indicate more favorable attitudes and greater knowledge.
Time Frame: 9-month follow-up, 18-month follow-up
Population: Analyses for the 9-month and 18-month follow-up visits include participants who had baseline data and completed the Parent Reading Belief Inventory (positive affect scale) at the 9-month and/or 18-month follow-up visit(s), respectively. Participants who did not participate in the 9-month follow-up were still welcome to participate in the 18-month follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual care including ROR | ROR plus text messages | ROR plus text messages plus connection to community resources
Number analyzed (Participants) | 181 | 176 | 187
score on a scale
  9-month follow-up: number analyzed (Participants) | 158 | 164 | 169
  9-month follow-up | 21.7 (3.9) | 21.6 (3.1) | 22.1 (3.3)
  18-month follow-up: number analyzed (Participants) | 168 | 168 | 172
  18-month follow-up | 20.1 (3.4) | 20.1 (2.9) | 19.8 (2.9)
Statistical Analysis 1: Comparison: Usual care including ROR vs ROR plus text messages; Analysis at the 9-month follow-up. A total of 630 parent-infant dyads (210 per arm) were needed to achieve 80% power to detect a 0.3 standard deviation (SD) difference assuming approximately 20% attrition. The null hypothesis was that there would be no differences between Arm 1 and Arm 2; Test type: Superiority; p = 0.80, ANOVA — The a priori threshold for statistical significance was p < .05
Statistical Analysis 2: Comparison: Usual care including ROR vs ROR plus text messages plus connection to community resources; Analysis at the 9-month follow-up. A total of 630 parent-infant dyads (210 per arm) were needed to achieve 80% power to detect a 0.3 standard deviation (SD) difference assuming approximately 20% attrition. The null hypothesis was that there would be no differences between Arm 1 and Arm 3; Test type: Superiority; p = 0.06, ANOVA — The a priori threshold for statistical significance was p < .05
Statistical Analysis 3: Comparison: Usual care including ROR vs ROR plus text messages; Analysis at the 18-month follow-up. \A total of 630 parent-infant dyads (210 per arm) were needed to achieve 80% power to detect a 0.3 standard deviation (SD) difference assuming approximately 20% attrition. The null hypothesis was that there would be no differences between Arm 1 and Arm 2; Test type: Superiority; p = 0.81, ANOVA — The a priori threshold for statistical significance was p < .05
Statistical Analysis 4: Comparison: Usual care including ROR vs ROR plus text messages plus connection to community resources; Analysis at the 18-month follow-up. A total of 630 parent-infant dyads (210 per arm) were needed to achieve 80% power to detect a 0.3 standard deviation (SD) difference assuming approximately 20% attrition. The null hypothesis was that there would be no differences between Arm 1 and Arm 3; Test type: Superiority; p = 0.08, ANOVA — The a priori threshold for statistical significance was p < .05

8. Secondary Outcome: Community Resource Participation
Description: Community resource participation was measured via the Survey of Income and Program Participation (SIPP), a series of questions that asks about caregiver and child participation in different types of community resources (e.g. food/nutrition support, income support, childcare assistance, etc.). Possible scores range from 0 to 17, with higher scores indicating more involvement in community resources.
Time Frame: Baseline, 9-month follow-up, 18-month follow-up
Population: Analyses for the 9-month and 18-month follow-up visits include participants who had baseline data and completed the SIPP at the 9-month and/or 18-month follow-up visit(s), respectively. Participants who did not participate in the 9-month follow-up were still welcome to participate in the 18-month follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual care including ROR | ROR plus text messages | ROR plus text messages plus connection to community resources
Number analyzed (Participants) | 209 | 210 | 211
score on a scale
  Baseline | 2.6 (1.2) | 2.5 (1.2) | 2.7 (1.2)
  9-month follow-up: number analyzed (Participants) | 166 | 170 | 178
  9-month follow-up | 2.4 (1.2) | 2.3 (1.1) | 2.5 (1.2)
  18-month follow-up: number analyzed (Participants) | 169 | 168 | 177
  18-month follow-up | 2.4 (1.0) | 2.4 (1.0) | 2.5 (1.1)
Statistical Analysis 1: Comparison: Usual care including ROR vs ROR plus text messages; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.07, ANOVA — The a priori threshold for statistical significance was p < .05
Statistical Analysis 2: Comparison: Usual care including ROR vs ROR plus text messages plus connection to community resources; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = 0.91, ANOVA — The a priori threshold for statistical significance was p < .05
Statistical Analysis 3: Comparison: Usual care including ROR vs ROR plus text messages; Analysis at the18-month follow-up. A total of 630 parent-infant dyads (210 per arm) were needed to achieve 80% power to detect a 0.3 standard deviation (SD) difference assuming approximately 20% attrition. The null hypothesis was that there would be no differences between Arm 1 and Arm 2; Test type: Superiority; p = 0.39, ANOVA — The a priori threshold for statistical significance was p < .05
Statistical Analysis 4: Comparison: Usual care including ROR vs ROR plus text messages plus connection to community resources; Analysis at the 18-month follow-up. \A total of 630 parent-infant dyads (210 per arm) were needed to achieve 80% power to detect a 0.3 standard deviation (SD) difference assuming approximately 20% attrition. The null hypothesis was that there would be no differences between Arm 1 and Arm 3; Test type: Superiority; p = 0.10, ANOVA — The a priori threshold for statistical significance was p < .05

9. Secondary Outcome: Caregiver-clinician Relationship
Description: The Physician-Parent Communication Survey is a caregiver reported measure of the caregiver-clinician relationship. We analyzed the interest subscale. The interest subscale includes 6 items are scored from 1 to 8. Scores from each item are averaged; thus total possible scores range from 1-8, with higher scores indicating stronger relationships.
Time Frame: Baseline; 9-month follow-up, 18-month follow-up
Population: Analyses for the 9-month and 18-month follow-up visits include participants who had baseline data and completed the Physician-Parent Communication Survey at the 9-month and/or 18-month follow-up visit(s), respectively. Participants who did not participate in the 9-month follow-up were still welcome to participate in the 18-month follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual care including ROR | ROR plus text messages | ROR plus text messages plus connection to community resources
Number analyzed (Participants) | 206 | 210 | 210
score on a scale
  Baseline | 5.8 (1.9) | 5.7 (1.9) | 5.5 (2.1)
  9-month follow-up: number analyzed (Participants) | 168 | 168 | 177
  9-month follow-up | 5.3 (2.0) | 5.3 (2.1) | 5.4 (2.0)
  18-month follow-up: number analyzed (Participants) | 168 | 168 | 176
  18-month follow-up | 4.9 (2.1) | 5.1 (2.1) | 4.8 (2.1)
Statistical Analysis 1: Comparison: Usual care including ROR vs ROR plus text messages; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.19, ANOVA — The a priori threshold for statistical significance was p < .05
Statistical Analysis 2: Comparison: Usual care including ROR vs ROR plus text messages plus connection to community resources; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = 0.18, ANOVA — The a priori threshold for statistical significance was p < .05
Statistical Analysis 3: Comparison: Usual care including ROR vs ROR plus text messages; Analysis at the 18-month follow-up. A total of 630 parent-infant dyads (210 per arm) were needed to achieve 80% power to detect a 0.3 standard deviation (SD) difference assuming approximately 20% attrition. The null hypothesis was that there would be no differences between Arm 1 and Arm 2; Test type: Superiority; p = 0.18, ANOVA — The a priori threshold for statistical significance was p < .05
Statistical Analysis 4: Comparison: Usual care including ROR vs ROR plus text messages plus connection to community resources; [analysis description as in outcome 7, analysis 4]; Test type: Superiority; p = 0.45, ANOVA — The a priori threshold for statistical significance was p < .05

10. Secondary Outcome: Social Needs and Stress
Description: Caregiver report of social needs and stressors was assessed via the Local Inventory of Needs and Knowledge (LINK) survey. Caregivers rate statements on social needs and stress from 0 to 4 with higher scores indicating greater needs and stress. Possible scores range from 0 to 16 with higher scores indicating greater needs and economic stress.
Time Frame: Baseline, 9-month follow-up, 18-month follow-up
Population: Analyses for the 9-month and 18-month follow-up visits include participants who had baseline data and completed the LINK at the 9-month and/or 18-month follow-up visit(s), respectively. Participants who did not participate in the 9-month follow-up were still welcome to participate in the 18-month follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual care including ROR | ROR plus text messages | ROR plus text messages plus connection to community resources
Number analyzed (Participants) | 204 | 203 | 206
score on a scale
  Baseline | 2.6 (1.1) | 2.7 (2.0) | 2.7 (1.1)
  9-month follow-up: number analyzed (Participants) | 166 | 165 | 176
  9-month follow-up | 2.8 (1.2) | 2.6 (1.2) | 2.8 (1.2)
  18-month follow-up: number analyzed (Participants) | 167 | 165 | 177
  18-month follow-up | 2.8 (1.2) | 2.7 (1.2) | 2.9 (1.2)
Statistical Analysis 1: Comparison: Usual care including ROR vs ROR plus text messages; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < .001, ANOVA — The a priori threshold for statistical significance was p < .05
Statistical Analysis 2: Comparison: Usual care including ROR vs ROR plus text messages plus connection to community resources; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = 0.68, ANOVA — The a priori threshold for statistical significance was p < .05
Statistical Analysis 3: Comparison: Usual care including ROR vs ROR plus text messages; [analysis description as in outcome 9, analysis 3]; Test type: Superiority; p = 0.16, ANOVA — The a priori threshold for statistical significance was p < .05
Statistical Analysis 4: Comparison: Usual care including ROR vs ROR plus text messages plus connection to community resources; [analysis description as in outcome 7, analysis 4]; Test type: Superiority; p = 0.39, ANOVA — The a priori threshold for statistical significance was p < .05

11. Secondary Outcome: Parent Stress
Description: The Parental Stress Scale is an eighteen-item measure that assesses parental stress. Scores range from 18 to 90 with higher scores indicating greater stress.
Time Frame: Baseline, 9-month follow-up, 18-month follow-up
Population: Analyses for the 9-month and 18-month follow-up visits include participants who had baseline data and completed the Parental Stress Scale at the 9-month and/or 18-month follow-up visit(s), respectively. Participants who did not participate in the 9-month follow-up were still welcome to participate in the 18-month follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual care including ROR | ROR plus text messages | ROR plus text messages plus connection to community resources
Number analyzed (Participants) | 200 | 206 | 207
score on a scale
  Baseline | 34.4 (7.9) | 35.1 (7.8) | 34.8 (7.5)
  9-month follow-up: number analyzed (Participants) | 166 | 171 | 178
  9-month follow-up | 34.9 (7.7) | 35.8 (8.6) | 34.7 (8.0)
  18-month follow-up: number analyzed (Participants) | 169 | 167 | 176
  18-month follow-up | 34.9 (7.5) | 34.5 (8.4) | 34.9 (7.6)
Statistical Analysis 1: Comparison: Usual care including ROR vs ROR plus text messages; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.87, ANOVA — The a priori threshold for statistical significance was p < .05
Statistical Analysis 2: Comparison: Usual care including ROR vs ROR plus text messages plus connection to community resources; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = 0.14, ANOVA — The a priori threshold for statistical significance was p < .05
Statistical Analysis 3: Comparison: Usual care including ROR vs ROR plus text messages; [analysis description as in outcome 9, analysis 3]; Test type: Superiority; p = 0.007, ANOVA — The a priori threshold for statistical significance was p < .05
Statistical Analysis 4: Comparison: Usual care including ROR vs ROR plus text messages plus connection to community resources; [analysis description as in outcome 7, analysis 4]; Test type: Superiority; p = 0.34, ANOVA — The a priori threshold for statistical significance was p < .05

12. Secondary Outcome: Child Media Use
Description: The ScreenQ is a caregiver report measure of media use in children. Scores range from 0 to 26 with higher score indicating more media use.
Time Frame: Baseline, 9-month follow-up, 18-month follow-up
Population: Analyses for the 9-month and 18-month follow-up visits include participants who had baseline data and completed the ScreenQ at the 9-month and/or 18-month follow-up visit(s), respectively. Participants who did not participate in the 9-month follow-up were still welcome to participate in the 18-month follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual care including ROR | ROR plus text messages | ROR plus text messages plus connection to community resources
Number analyzed (Participants) | 209 | 210 | 211
score on a scale
  Baseline | 4.9 (3.2) | 4.7 (2.7) | 4.6 (2.9)
  9-month follow-up: number analyzed (Participants) | 168 | 171 | 178
  9-month follow-up | 5.2 (2.6) | 5.1 (2.7) | 4.9 (2.6)
  18-month follow-up: number analyzed (Participants) | 169 | 168 | 178
  18-month follow-up | 5.2 (2.2) | 5.1 (2.3) | 4.9 (2.2)
Statistical Analysis 1: Comparison: Usual care including ROR vs ROR plus text messages; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.99, ANOVA — The a priori threshold for statistical significance was p < .05
Statistical Analysis 2: Comparison: Usual care including ROR vs ROR plus text messages plus connection to community resources; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = 0.07, ANOVA — The a priori threshold for statistical significance was p < .05
Statistical Analysis 3: Comparison: Usual care including ROR vs ROR plus text messages; [analysis description as in outcome 9, analysis 3]; Test type: Superiority; p = 0.41, ANOVA — The a priori threshold for statistical significance was p < .05
Statistical Analysis 4: Comparison: Usual care including ROR vs ROR plus text messages plus connection to community resources; [analysis description as in outcome 7, analysis 4]; Test type: Superiority; p = 0.03, ANOVA — The a priori threshold for statistical significance was p < .05

13. Other Pre Specified Outcome: ROR Receipt
Description: Caregiver's report of receipt of literacy promotion components during their previous healthcare visit.
Time Frame: Baseline; 9-month follow up; 18-month follow up
Population: Analyses for the 9-month and 18-month follow-up visits include participants who had baseline data and completed the 9-month and/or 18-month follow-up visit(s), respectively. Participants who did not participate in the 9-month follow-up were still welcome to participate in the 18-month follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual care including ROR | ROR plus text messages | ROR plus text messages plus connection to community resources
Number analyzed (Participants) | 209 | 210 | 211
Participants
  Baseline 0 components | 51 | 57 | 63
  Baseline 1 component | 52 | 53 | 42
  Baseline 2 components | 73 | 73 | 72
  Baseline 3 components | 33 | 27 | 34
  9-month follow-up 0 componenets: number analyzed (Participants) | 168 | 173 | 178
  9-month follow-up 0 componenets | 64 | 57 | 56
  9-month follow up 1 component: number analyzed (Participants) | 168 | 173 | 178
  9-month follow up 1 component | 36 | 40 | 48
  9-month follow-up 2 components: number analyzed (Participants) | 168 | 173 | 178
  9-month follow-up 2 components | 45 | 52 | 46
  9-month follow-up 3 components: number analyzed (Participants) | 168 | 173 | 178
  9-month follow-up 3 components | 23 | 24 | 28
  18-month follow-up 0 components: number analyzed (Participants) | 170 | 169 | 178
  18-month follow-up 0 components | 70 | 51 | 61
  18-month follow-up 1 component: number analyzed (Participants) | 170 | 169 | 178
  18-month follow-up 1 component | 31 | 50 | 51
  18-month follow-up 2 components: number analyzed (Participants) | 170 | 169 | 178
  18-month follow-up 2 components | 45 | 36 | 42
  18-month follow-up 3 components: number analyzed (Participants) | 170 | 169 | 178
  18-month follow-up 3 components | 24 | 32 | 24

14. Other Pre Specified Outcome: Observed Parent-child Interactions
Description: Observation of parent-child interactions during shared reading and free play; observations will be coded based on DialogPR items
Time Frame: 9-month follow up
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Deaths, serious adverse events, and other (non-serious adverse events) were not assessed for study participants.
Arm/Group | Usual care including ROR | ROR plus text messages | ROR plus text messages plus connection to community resources
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-14): https://cdn.clinicaltrials.gov/large-docs/53/NCT04609553/Prot_SAP_001.pdf
  • Informed Consent Form (2024-10-14): https://cdn.clinicaltrials.gov/large-docs/53/NCT04609553/ICF_000.pdf